CLINICAL TRIAL: NCT07335198
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Efimosfermin Alfa Administered as a Single Dose to Healthy Participants of Chinese, Japanese, and White/European Ancestry
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Efimosfermin Alfa Administered as a Single Dose to Healthy Participants of Chinese, Japanese, and White/European Ancestry
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 301158
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Efimosfermin alfa; Placebo; First time in Asia; Chinese; Japanese; White/Europeans; Pharmacokinetics; Safety
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Efimosfermin alfa in participants of Chinese Ancestry (Experimental): Healthy participants of Chinese ancestry will be randomized to receive efimosfermin alfa.
  Interventions: Drug: Efimosfermin alfa
- Efimosfermin alfa in participants of Japanese Ancestry (Experimental): Healthy participants of Japanese ancestry will be randomized to receive efimosfermin alfa.
  Interventions: Drug: Efimosfermin alfa
- Efimosfermin alfa in participants of White/European Ancestry (Experimental): Healthy participants of White/European ancestry will be randomized to receive efimosfermin alfa
  Interventions: Drug: Efimosfermin alfa
- Placebo in participants of Chinese Ancestry (Placebo Comparator): Healthy participants of Chinese ancestry will be randomized to receive Placebo.
  Interventions: Drug: Placebo
- Placebo in participants of Japanese Ancestry (Placebo Comparator): Healthy participants of Japanese ancestry will be randomized to receive Placebo.
  Interventions: Drug: Placebo
- Placebo in participants of White/European Ancestry (Placebo Comparator): Healthy participants of White/European ancestry will be randomized to receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efimosfermin alfa — Efimosfermin alfa to be administered
  Arms: Efimosfermin alfa in participants of Chinese Ancestry; Efimosfermin alfa in participants of Japanese Ancestry; Efimosfermin alfa in participants of White/European Ancestry
Drug: Placebo — Placebo to be administered
  Arms: Placebo in participants of Chinese Ancestry; Placebo in participants of Japanese Ancestry; Placebo in participants of White/European Ancestry

SUMMARY:
This is a first time in Asia (FTIA) study designed to evaluate the safety, tolerability, pharmacokinetic (PK) and immunogenicity of efimosfermin alfa to healthy participants of Chinese, Japanese, and White/European ancestry.

ELIGIBILITY:
Inclusion Criteria:

Participants who are generally healthy as determined by medical evaluation

* Body weight at least 50.0 Kilogram (kg) for male participants or at least 45.0 kg for female participants
* Body mass index (BMI) within the range of 18.0 to 28.0 kilograms per square meter (kg/m^2) (inclusive)
* Male and female participants
* Participants of Chinese ancestry are eligible if born in mainland China, Hong Kong, or Taiwan, and have lived outside China, Hong Kong, or Taiwan for less than 10 years at the time of screening.
* Participants of Japanese ancestry are eligible if born in Japan and Descendant of 2 ethnic Japanese parents and 4 ethnic Japanese grandparents; and. have lived outside Japan for less than 10 years at the time of screening.
* Participants of White/European ancestry are eligible if self-identified as being of White/European ancestry, (i.e., from the original peoples of Europe) irrespective of current place of residence; and.
* Descendant of 2 parents and 4 grandparents of White/European ancestry (that is [i.e.], from the original peoples of Europe) irrespective of place of birth or current place of residence.

Exclusion Criteria:

* History or presence of disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Current or chronic history of liver or biliary disease with the exception of Gilbert's syndrome or asymptomatic gallstones.
* History of pancreatic injury, pancreatitis or other pancreatic disease; history of Type one Diabetes Mellitus (T1DM) or positive glutamic acid decarboxylase auto-antibodies, or major Type two Diabetes Mellitus (T2DM) complications including severe gastroparesis and autonomic neuropathy.
* Abnormal blood pressure (defined as systolic Blood Pressure (BP) more than equal (>=)140 millimeters of mercury (mmHg) or diastolic BP >=90 mmHg) measured based on the average of triplicate BP readings).
* History of metabolic bone disorders including osteoporosis, osteopenia, or osteomalacia.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
* Alanine transaminase (ALT) more than (>)1.5 * upper limit of normal (ULN).
* Total bilirubin >1.5 * ULN
* Known bleeding disorder.
* History of immunodeficiency diseases, including a positive test result for human immunodeficiency virus (HIV).
* Corrected QT Interval using Fridericia's Formula. (QTcF) >=450 millisecond (msec)(male) or >=470 msec (female) at Screening Visit based on the average of triplicate ECGs.
* Use of statins, other lipid lowering medications or hypertension medications unless on a stable dose for at least 3 months.
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days, whichever was longer; or longer if required by local regulations.
* Participants who have received native FGF21 or a FGF21 analog at any time in the past.
* Intended use of over the counter (OTC) or prescription medication (including herbal medications) within 7 days prior to dosing and for the duration of study participation.
* Live vaccine within 14 days prior to dosing and non-live vaccines for 7 days prior study dosing.
* Current enrolment or participation in another clinical trial within the last 30 days before signing consent of current study.
* Presence of hepatitis B surface antigen (HBsAg) or hepatitis C antibody at screening or within 3 months prior to the first dose of study intervention
* A positive pre-study drug/alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs), treatment related AEs and serious adverse events (SAEs) | Up to 90 days
Number of participants with clinically significant changes in hematology, chemistry and urinalysis parameters | Up to 90 days
Number of participants with clinically significant changes in 12 Lead electrocardiogram (ECG) | Up to 90 days
Number of participants with clinically significant changes in vital signs | Up to 90 days
Area under the serum drug concentration versus time curve from time zero to the time of the last quantifiable concentration (AUC[0-t]) of efimosfermin alfa | Up to 90 days
Area under the serum drug concentration versus time curve from time zero extrapolated to infinity (AUC[0-inf]) of efimosfermin alfa | Up to 90 days
Maximum observed serum drug concentration, determined directly from the serum concentration-time data (Cmax) of efimosfermin alfa | Up to 90 days

SECONDARY OUTCOMES:
Time to maximum observed serum drug concentration (Tmax) of efimosfermin alfa | Up to 90 days
Apparent terminal phase half-life (t1/2) of efimosfermin alfa | Up to 90 days
Area under the serum drug concentration versus time curve from time zero to 90 days [AUC(0-90days)] of efimosfermin alfa | Up to 90 days
Time of last quantifiable plasma drug concentration (Tlast) of efimosfermin alfa | Up to 90 days
Apparent clearance (CL/F) of efimosfermin alfa | Up to 90 days
Apparent volume of distribution (Vz/F) of efimosfermin alfa | Up to 90 days
Apparent terminal phase elimination rate constant (Lambda_z) of efimosfermin alfa | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf